CLINICAL TRIAL: NCT01727544
Title: Objective Assessment of Vestibular Function Outcome After Cartilage Cap Occlusion Surgery for Dehiscent Superior Semicircular Canal
Brief Title: Vestibular Function Outcome After Cartilage Cap Occlusion Surgery
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Changed to a retrospective chart review
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Larry B. Lundy, PI, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-001953
Record Dates: First submitted 2012-08-22; First posted 2012-11-16 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Vestibular Dizziness; Superior Semicircular Canal Dehiscence
Keywords: superior semicircular canal; non-vestibular dizziness; vestibular dizziness
MeSH Terms: conditions — Semicircular Canal Dehiscence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgical Group (Active Comparator): patients will undergo a primary transmastoid and tegmen mini-craniotomy cartilage cap occlusion surgery.
  Interventions: Procedure: cartilage cap occlusion surgery
- Non Surgical Group (No Intervention): patients meet the same criteria but will elect not to undergo surgery

INTERVENTIONS:
Procedure: cartilage cap occlusion surgery — placement of a cartilage cap over the dome of the superior semicircular canal through a combined transmastoid and tegmen mini- craniotomy approach.
  Arms: Surgical Group

SUMMARY:
The primary objective of this study is to measure objective, functional outcomes of patients undergoing cartilage cap occlusion surgery for a dehiscent superior semicircular canal.

DETAILED DESCRIPTION:
One option for managing a dehiscent superior semicircular canal is surgical intervention. One of the surgical techniques is the transmastoid and tegmen mini-craniotomy cartilage cap occlusion of the dehiscent superior semicircular canal.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory
* independent self-sufficient adults
* good general health
* medically stable

Exclusion Criteria:

* Medically unstable
* pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
objective improvement | baseline to 3 months
  The primary outcome measure will be the subsequent (3 month) FGA scores between the control group and the surgery group to assess any objective improvement attributable to surgery

SECONDARY OUTCOMES:
ABC Scale | baseline to 3 months
  Secondary objective outcome measures will be changes in conductive hearing loss and changes in cervical VEMP thresholds between the two groups at the 3-month interval. Secondary subjective outcome measures will be ABC Scale and VAS scores between the two groups at 3 months.
VAS scores | baseline to 3 months
  Secondary objective outcome measures will be changes in conductive hearing loss and changes in cervical VEMP thresholds between the two groups at the 3-month interval. Secondary subjective outcome measures will be ABC Scale and VAS scores between the two groups at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Larry Lundy, MD, Principal Investigator — Mayo Clinic